CLINICAL TRIAL: NCT04123834
Title: Functional Outcome Comparison of Implant-Free Bone-Patellar Tendon Autografts Using Press-Fit Fixation Technique and Hamstring Autografts Using Implant in Arthroscopic Anterior Cruciate Ligament Reconstruction: A Prospective Study
Brief Title: Functional Outcome Comparison of Implant-Free Bone-Patellar Tendon Autograft in Arthroscopic ACL Reconstruction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Andri Maruli Tua Lubis, Principal Investigator, Indonesia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Press-Fit ACL
Record Dates: First submitted 2019-09-29; First posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Anterior Cruciate Ligament Injuries; Ligament; Rupture, Knee, Spontaneous; Tendon Graft; Complication, Mechanical
Keywords: anterior cruciate ligament; anterior cruciate ligament injury; implantless ACL reconstruction; press-fit fixation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Rupture

STUDY DESIGN:
Intervention Model Description: A prospective cohort study design was used. Between March 2013 and March 2014, 12 patients underwent implantless ACL reconstruction using press-fit femoral technique, while 24 patients underwent implant ACL reconstruction. Objective functional outcome were measured using rolimeter, and subjective functional outcome were measured according to IKDC, Tegner-Lysholm and KOOS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- implantless Arthroscopic ACL reconstruction (Experimental): implantless Arthroscopic ACL reconstruction using press-fit femoral technique
  Interventions: Procedure: Patella tendon & bone block autograft + press-fit femoral technique; Procedure: Arthroscopic ACL reconstruction
- Arthroscopic ACL reconstruction with implant (Experimental): ACL reconstruction with implant (hamstring autograft fixed with bioscrew and endo-button)
  Interventions: Procedure: Arthroscopic ACL reconstruction; Device: Hamstring tendon autograft + implant fixation

INTERVENTIONS:
Procedure: Patella tendon & bone block autograft + press-fit femoral technique — Implantless Arthroscopic ACL reconstruction using press-fit femoral technique The investigator's study uses the press-fit graft fixation technique by Edgar Michael. A midline skin incision was made that extends from inferior pole of patella up to anterior tibial tuberosity. Patella tendon with tibial tuberosity bone block were harvested, patella bone was left intact. The tendon was fixed together with non-absorbable suture.
  Arms: implantless Arthroscopic ACL reconstruction
Procedure: Arthroscopic ACL reconstruction — Arthroscopic ACL reconstruction with implant (using hamstring autograft fixed with bioscrew and endo-button)
Device: Hamstring tendon autograft + implant fixation — Arthroscopic ACL reconstruction with implant (using hamstring tendon autograft fixed with bioscrew and endo-button)
  Arms: Arthroscopic ACL reconstruction with implant

SUMMARY:
The use of implants for conventional anterior cruciate ligament (ACL) graft fixation has been associated with several problems including graft injury, implant osteolysis, implant migration and soft tissue irritation. Implantless ACL surgery offers additional benefits involving lower cost, improved graft incorporation and ease of revision surgery. The investigators aimed to compare the functional outcome of implantless bone-patellar tendon autograft using press-fit fixation technique and hamstring autografts using implant.

DETAILED DESCRIPTION:
Purpose: The use of implants for conventional anterior cruciate ligament (ACL) graft fixation has been associated with several problems including graft injury, implant osteolysis, implant migration and soft tissue irritation. Implantless ACL surgery offers additional benefits involving lower cost, improved graft incorporation and ease of revision surgery. The investigators aimed to compare the functional outcome of implantless bone-patellar tendon autograft using press-fit fixation technique and hamstring autografts using implant.

Materials and Methods: A prospective cohort study design was used. Between March 2013 and March 2014, 12 patients underwent implantless ACL reconstruction using press-fit femoral technique, while 24 patients underwent implant ACL reconstruction. Objective functional outcome were measured using rolimeter, and subjective functional outcome were measured according to IKDC, Tegner-Lysholm and KOOS.

ELIGIBILITY:
Inclusion Criteria:

* total rupture of ACL on a single knee

Exclusion Criteria:

* increased knee laxity according to Beighton Hypermobility Score
* previous history of knee surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2014-03-30 (Actual); Study Completion 2014-03-30 (Actual)

PRIMARY OUTCOMES:
Anterior knee laxity | At 1 month after surgery.
  Anterior knee laxity (in centimetres) was assessed by measuring anterior translation at 30° of flexion with a rolimeter and comparing it with the contralateral knee.
Anterior knee laxity | At 3 months after surgery.
  Anterior knee laxity (in centimetres) was assessed by measuring anterior translation at 30° of flexion with a rolimeter and comparing it with the contralateral knee.
Anterior knee laxity | At 6 months after surgery.
  Anterior knee laxity (in centimetres) was assessed by measuring anterior translation at 30° of flexion with a rolimeter and comparing it with the contralateral knee.
Functional outcome score International Knee Documentation committee (IKDC) | At 1 month after surgery.
  International Knee Documentation committee (IKDC) score evaluate improvement or deterioration in symptoms, function, and sports activities.
  Number of items: 18 subscales:
  * symptoms: pain, stiffness, swelling, locking/catching and giving-way of the knee.
  * sports activities: functions such as going up and down the stairs, rising from a chair, squatting and jumping
  * function and activity of daily living: knee condition prior to injury
  Response options vary for each item. Item 6 dichotomizes response into yes/no; items 1, 4, 5, 7, 8, and 9 use 5-point Likert scales; and items 2, 3, and 10 use 11-point numerical rating scales. The total score is calculated as (sum of items)/(maximum possible score) × 100. Possible score range 0-100, where 100 = no limitation with daily or sporting activities and the absence of symptoms. Higher values represent a better outcome.
Functional outcome score International Knee Documentation committee (IKDC) | At 3 months after surgery.
  International Knee Documentation committee (IKDC) score evaluate improvement or deterioration in symptoms, function, and sports activities.
  Number of items: 18 subscales:
  * symptoms: pain, stiffness, swelling, locking/catching and giving-way of the knee.
  * sports activities: functions such as going up and down the stairs, rising from a chair, squatting and jumping
  * function and activity of daily living: knee condition prior to injury
  Response options vary for each item. Item 6 dichotomizes response into yes/no; items 1, 4, 5, 7, 8, and 9 use 5-point Likert scales; and items 2, 3, and 10 use 11-point numerical rating scales. The total score is calculated as (sum of items)/(maximum possible score) × 100. Possible score range 0-100, where 100 = no limitation with daily or sporting activities and the absence of symptoms. Higher values represent a better outcome.
Functional outcome score International Knee Documentation committee (IKDC) | At 6 months after surgery.
  International Knee Documentation committee (IKDC) score evaluate improvement or deterioration in symptoms, function, and sports activities.
  Number of items: 18 subscales:
  * symptoms: pain, stiffness, swelling, locking/catching and giving-way of the knee.
  * sports activities: functions such as going up and down the stairs, rising from a chair, squatting and jumping
  * function and activity of daily living: knee condition prior to injury
  Response options vary for each item. Item 6 dichotomizes response into yes/no; items 1, 4, 5, 7, 8, and 9 use 5-point Likert scales; and items 2, 3, and 10 use 11-point numerical rating scales. The total score is calculated as (sum of items)/(maximum possible score) × 100. Possible score range 0-100, where 100 = no limitation with daily or sporting activities and the absence of symptoms. Higher values represent a better outcome.
Functional outcome score Tegner-Lysholm | At 1 month after surgery.
  Tegner-Lysholm Score subjectively evaluate to how the knee pain has affected the ability to manage in everyday life.
  Number of items: 8 items, each scored differently
  Subscales:
  1. limp (0, 3, 5)
  2. support (0, 2, 5)
  3. locking (0, 2, 6, 10, 15)
  4. instability (0, 5, 10, 15, 20, 25)
  5. pain (0, 5, 10, 15, 20, 25)
  6. swelling (0, 2, 6, 10)
  7. stair climbing (0, 2, 6, 10)
  8. squatting (0, 2, 4, 5)
  Total score is given as "excellent" for 95 to 100 points; "good" for 84 to 94 points, "fair" for 65 to 83 points, or "poor" for less than 65 points.
Functional outcome scores Tegner-Lysholm | At 3 months after surgery.
  Tegner-Lysholm Score subjectively evaluate to how the knee pain has affected the ability to manage in everyday life.
  Number of items: 8 items, each scored differently
  Subscales:
  1. limp (0, 3, 5)
  2. support (0, 2, 5)
  3. locking (0, 2, 6, 10, 15)
  4. instability (0, 5, 10, 15, 20, 25)
  5. pain (0, 5, 10, 15, 20, 25)
  6. swelling (0, 2, 6, 10)
  7. stair climbing (0, 2, 6, 10)
  8. squatting (0, 2, 4, 5)
  Total score is given as "excellent" for 95 to 100 points; "good" for 84 to 94 points, "fair" for 65 to 83 points, or "poor" for less than 65 points.
Functional outcome scores Tegner-Lysholm | At 6 months after surgery.
  Tegner-Lysholm Score subjectively evaluate to how the knee pain has affected the ability to manage in everyday life.
  Number of items: 8 items, each scored differently
  Subscales:
  1. limp (0, 3, 5)
  2. support (0, 2, 5)
  3. locking (0, 2, 6, 10, 15)
  4. instability (0, 5, 10, 15, 20, 25)
  5. pain (0, 5, 10, 15, 20, 25)
  6. swelling (0, 2, 6, 10)
  7. stair climbing (0, 2, 6, 10)
  8. squatting (0, 2, 4, 5)
  Total score is given as "excellent" for 95 to 100 points; "good" for 84 to 94 points, "fair" for 65 to 83 points, or "poor" for less than 65 points.
Functional outcome score Knee Injury and Osteoarthritis Outcome (KOOS) | At 1 month after surgery.
  Knee Injury and Osteoarthritis Outcome (KOOS) measure patients' opinions about their knee and associated problems over short- and long-term followup (1 week to decades).
  Number of items: 42 items rated on a 5-point Likert scale (0-4) across 5 subscales:
  * pain frequency and severity during functional activities (subscale score range: 0-36)
  * symptoms such as the severity of knee stiffness and the presence of swelling, grinding or clicking, catching, and range of motion restriction (subscale score range: 0-28)
  * difficulty experienced during activities of daily living (ADL) (subscale score range: 0-68)
  * difficulty experienced with sport and recreational activities (subscale score range: 0-20)
  * knee-related quality of life (QOL) (subscale score range: 0-16)
  The 5 dimensions are scored separately as the sum of all corresponding items, and then converted into percentage (score range 0-100). Score of 0 means extreme knee problems and score of 100 means no knee problems.
Functional outcome score Knee Injury and Osteoarthritis Outcome (KOOS) | At 3 months after surgery.
  Knee Injury and Osteoarthritis Outcome (KOOS) measure patients' opinions about their knee and associated problems over short- and long-term followup (1 week to decades).
  Number of items: 42 items rated on a 5-point Likert scale (0-4) across 5 subscales:
  * pain frequency and severity during functional activities (subscale score range: 0-36)
  * symptoms such as the severity of knee stiffness and the presence of swelling, grinding or clicking, catching, and range of motion restriction (subscale score range: 0-28)
  * difficulty experienced during activities of daily living (ADL) (subscale score range: 0-68)
  * difficulty experienced with sport and recreational activities (subscale score range: 0-20)
  * knee-related quality of life (QOL) (subscale score range: 0-16)
  The 5 dimensions are scored separately as the sum of all corresponding items, and then converted into percentage (score range 0-100). Score of 0 means extreme knee problems and score of 100 means no knee problems.
Functional outcome score Knee Injury and Osteoarthritis Outcome (KOOS) | At 6 months after surgery.
  Knee Injury and Osteoarthritis Outcome (KOOS) measure patients' opinions about their knee and associated problems over short- and long-term followup (1 week to decades).
  Number of items: 42 items rated on a 5-point Likert scale (0-4) across 5 subscales:
  * pain frequency and severity during functional activities (subscale score range: 0-36)
  * symptoms such as the severity of knee stiffness and the presence of swelling, grinding or clicking, catching, and range of motion restriction (subscale score range: 0-28)
  * difficulty experienced during activities of daily living (ADL) (subscale score range: 0-68)
  * difficulty experienced with sport and recreational activities (subscale score range: 0-20)
  * knee-related quality of life (QOL) (subscale score range: 0-16)
  The 5 dimensions are scored separately as the sum of all corresponding items, and then converted into percentage (score range 0-100). Score of 0 means extreme knee problems and score of 100 means no knee problems.

CONTACTS AND LOCATIONS:
Overall Officials: Andri MT Lubis, MD, PhD, Principal Investigator — Indonesia University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biau DJ, Tournoux C, Katsahian S, Schranz PJ, Nizard RS. Bone-patellar tendon-bone autografts versus hamstring autografts for reconstruction of anterior cruciate ligament: meta-analysis. BMJ. 2006 Apr 29;332(7548):995-1001. doi: 10.1136/bmj.38784.384109.2F. Epub 2006 Apr 7. PMID 16603564
- [Background] Frobell RB, Roos EM, Roos HP, Ranstam J, Lohmander LS. A randomized trial of treatment for acute anterior cruciate ligament tears. N Engl J Med. 2010 Jul 22;363(4):331-42. doi: 10.1056/NEJMoa0907797. PMID 20660401
- [Background] Romanini E, D'Angelo F, De Masi S, Adriani E, Magaletti M, Lacorte E, Laricchiuta P, Sagliocca L, Morciano C, Mele A. Graft selection in arthroscopic anterior cruciate ligament reconstruction. J Orthop Traumatol. 2010 Dec;11(4):211-9. doi: 10.1007/s10195-010-0124-9. Epub 2010 Dec 23. PMID 21181226
- [Background] Remer EM, Fitzgerald SW, Friedman H, Rogers LF, Hendrix RW, Schafer MF. Anterior cruciate ligament injury: MR imaging diagnosis and patterns of injury. Radiographics. 1992 Sep;12(5):901-15. doi: 10.1148/radiographics.12.5.1529133.
- [Background] Tirmik U, Mahirogullari M, Kuskucu M. The results of reconstruction of the ACL using the cross-pin femoral system and four-strand hamstring tendon autografts. Acta Orthop Traumatol Turc. 2011;45(4):233-9. doi: 10.3944/AOTT.2011.2309. PMID 21908962
- [Background] Mei Y, Ao YF, Wang JQ, Ma Y, Zhang X, Wang JN, Zhu JX. Clinical characteristics of 4355 patients with anterior cruciate ligament injury. Chin Med J (Engl). 2013 Dec;126(23):4487-92. PMID 24286412
- [Background] Taketomi S, Inui H, Yamagami R, Shirakawa N, Kawaguchi K, Nakagawa T, Tanaka S. Bone-Patellar Tendon-Bone Autograft versus Hamstring Tendon Autograft for Anatomical Anterior Cruciate Ligament Reconstruction with Three-Dimensional Validation of Femoral and Tibial Tunnel Positions. J Knee Surg. 2018 Oct;31(9):866-874. doi: 10.1055/s-0037-1615813. Epub 2017 Dec 28. PMID 29284176
- [Background] Pavlik A, Hidas P, Tallay A, Toman J, Berkes I. Femoral press-fit fixation technique in anterior cruciate ligament reconstruction using bone-patellar tendon-bone graft: a prospective clinical evaluation of 285 patients. Am J Sports Med. 2006 Feb;34(2):220-5. doi: 10.1177/0363546505279920. Epub 2005 Oct 6. PMID 16210575
- [Background] Noyes FR, Barber-Westin SD. Treatment of meniscus tears during anterior cruciate ligament reconstruction. Arthroscopy. 2012 Jan;28(1):123-30. doi: 10.1016/j.arthro.2011.08.292. Epub 2011 Nov 9. PMID 22074619
- [Background] Widuchowski W, Widuchowska M, Koczy B, Dragan S, Czamara A, Tomaszewski W, Widuchowski J. Femoral press-fit fixation in ACL reconstruction using bone-patellar tendon-bone autograft: results at 15 years follow-up. BMC Musculoskelet Disord. 2012 Jun 27;13:115. doi: 10.1186/1471-2474-13-115. PMID 22738187
- [Background] Wipfler B, Donner S, Zechmann CM, Springer J, Siebold R, Paessler HH. Anterior cruciate ligament reconstruction using patellar tendon versus hamstring tendon: a prospective comparative study with 9-year follow-up. Arthroscopy. 2011 May;27(5):653-65. doi: 10.1016/j.arthro.2011.01.015. PMID 21663722

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-03-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT04123834/Prot_SAP_000.pdf
  • Informed Consent Form (2013-03-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT04123834/ICF_001.pdf